CLINICAL TRIAL: NCT06198569
Title: The Effect of Scapular Proprioceptive Neuromuscular Facilitation (PNF) Exercises on Posture, Upper Extremity Strength and Dexterity in University Students.
Brief Title: The Effect of Scapular Proprioceptive Neuromuscular Facilitation (PNF) Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Zekiye İpek KATIRCI KIRMACI, Asst. Prof, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZİKK
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Postural Kyphosis
Keywords: PNF; Scapular exercise
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): STRENGTH EXERCISE TRAINING
  Interventions: Other: strength exercises
- Study Group (Experimental): PNF EXERCISE TRAINING
  Interventions: Other: PNF EXERCISES

INTERVENTIONS:
Other: PNF EXERCISES — Scapular PNF exercise training (6 Weeks) Exercise Frequency 3 days/week Exercise Intensity 60% of 1 maximum repetition Exercise Duration: 5-minute warm-up 20 minutes (2 sets of 15 repetitions) exercise training 5 min cool down Exercise Type Scapular patterns
  * Anterior elevation-Posterior depression
  * Anterior depression-Posterior elevation PNF techniques
  * Repetitive stretching
  * Rhythmic stabilization
  Arms: Study Group
Other: strength exercises — Upper limb exercise training (6 Weeks) 3 days/week 60% of 1 repetition maximum 5 minute warm up 20 min exercise training 5 min cool down
  Upper extremity movements - Scapular retraction - Shoulder flexion - Shoulder extension - Shoulder abduction - Shoulder adduction Resistant exercise training with Theraband and weights
  Arms: Control Group

SUMMARY:
Posture is generally defined as the sitting or standing position of a person's body. Repetitive or prolonged positioning in an atypical posture may also occur as a risk factor for the development of musculoskeletal diseases. Race, gender, seasons, nutrition, socio-economic status, profession and occupations, psychological state, hygiene, sleep patterns, exercise habits, fatigue, fractures, soft tissue disorders, disorders in the normal alignment angles of the joints, and emotional states such as joy, grief, and distress. It affects posture. Creating professional awareness among physiotherapy and rehabilitation students is very important for the physiotherapy profession, which has a very important role in protecting and improving public health, to achieve its professional goals. On the other hand, physiotherapists and physiotherapy students are at great risk of musculoskeletal disorders due to their working conditions and working postures.

The basic principle of proprioceptive neuromuscular facilitation techniques, defined as facilitating the responses of the neuromuscular mechanism by stimulating the proprioceptors and briefly referred to as PNF, is based on the principle that physiological movements in the human body have rotational and oblique characters and that a greater response can be achieved with movements performed against maximum resistance. The shoulder girdle serves purposes beyond stabilization and movement of the extremities. The clavicle and scapula cooperate as a single unit in the shoulder girdle. The scapula is not a weight-bearing structure during normal functions; rather, it supports the attachment of skeletal muscles.

DETAILED DESCRIPTION:
Posture is generally defined as the sitting or standing position of a person's body. Repetitive or prolonged positioning in an atypical posture may also occur as a risk factor for the development of musculoskeletal diseases. Race, gender, seasons, nutrition, socio-economic status, profession and occupations, psychological state, hygiene, sleep patterns, exercise habits, fatigue, fractures, soft tissue disorders, disorders in the normal alignment angles of the joints, and emotional states such as joy, grief, and distress. It affects posture. Creating professional awareness among physiotherapy and rehabilitation students is very important for the physiotherapy profession, which has a very important role in protecting and improving public health, to achieve its professional goals. On the other hand, physiotherapists and physiotherapy students are at great risk of musculoskeletal disorders due to their working conditions and working postures.

The basic principle of proprioceptive neuromuscular facilitation techniques, defined as facilitating the responses of the neuromuscular mechanism by stimulating the proprioceptors and briefly referred to as PNF, is based on the principle that physiological movements in the human body have rotational and oblique characters and that a greater response can be achieved with movements performed against maximum resistance. The shoulder girdle serves purposes beyond stabilization and movement of the extremities. The clavicle and scapula cooperate as a single unit in the shoulder girdle. The scapula is not a weight-bearing structure during normal functions; rather, it supports the attachment of skeletal muscles.Scapula patterns are activated by upper extremity patterns, and all upper extremity patterns occur together with scapula patterns. The therapeutic purposes of scapula patterns are as follows:

mobility and stabilization of the scapula,

* Trunk muscles and movements, rotation, etc. functional activities,
* Cervical movements and stability, to increase upper-extremity movements and stabilization. Strengthening exercises for posture problems are frequently included in literature studies. However, the results of scapular-pattern PNF exercises specific to the shoulder girdle muscles are unknown. In this study, which we planned in light of this information, the findings obtained from scapular PNF exercises will serve to fill this gap in the literature.

Our hypotheses in this project are:

Hypothesis 1: Scapular PNF applications will show superiority in the development of muscle strength compared to upper extremity strengthening exercises in university students who receive 6-week training.

Hypothesis 2: Scapular PNF applications will be superior to upper extremity strengthening exercises in correcting shoulder girdle posture in university students who receive 6-week training.

Hypothesis 3: Scapular PNF applications will be superior to upper extremity strengthening exercises in the development of hand skills in university students who receive 6-week training.

The most common posture problem seen in university students is the deterioration of shoulder girdle posture. In this project,

1. Purpose: To examine the effects of scapular PNF training on the strength of upper extremity muscles.
2. Purpose: To examine the effects of scapular PNF training on shoulder girdle posture.

Purpose: To examine the effects of scapular PNF training on manual skills.

ELIGIBILITY:
Inclusion Criteria:

1. Being between the ages of 18-35
2. Volunteering to participate in the study

Exclusion Criteria:

1. Having a systemic disease that prevents exercise,
2. Having a history of orthopedic problems in the upper extremity (fracture, trauma, etc.)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | Baseline and after 6 weeks
  Lower extremity muscle strength will be measured with a digital muscle dynamometer. Lower extremity muscles will be evaluated using a digital dynamometer (Knect). With this device, muscle force values are expressed in Newton (N). Muscle strength will be recorded by making 3 measurements with a digital dynamometer, on the right and left extremities, without allowing the patients to compensate, and the average values will be used.
Posture | Baseline and after 6 weeks
  It will be done with the PostureScreen Mobile (PSM) application. Using the phone's camera application, participants will be photographed from 4 directions: front, back (coronal plane), right and left (sagittal plane). After the photo is taken, after marking the anatomical points specified in the application, the function of the application is started and the right or left shift and tilt angles of the head, shoulders, rib cage, hips from the front, the tilt angles of the head, shoulders, hips, knees from the side and the head, shoulders, rib cage from the back are displayed. , right and left tilt and shift angles of the midpoint of the hip, T1-T4, T4-T8, T8-T12, T12-L3 vertebrae, L3 and SIPS will be determined and recorded. The application is a valid and reliable method and its ICC score is between 0.71-0.99.
Manual skills | Baseline and after 6 weeks
  Will be evaluated with Purdue-Peg board test (PPBT). It is one of the tests frequently used in personnel selection for jobs requiring motor skills and coordination. It is a test that also measures the fingertip dexterity required for assembly work. Washers, rings and small nails are used in this test. The completion time of the test is recorded in seconds. The test is valid and reliable.

CONTACTS AND LOCATIONS:
Overall Officials: Zekiye İpek Katırcı Kırmacı, Principal Investigator — Gaziantep Islam Science and Technology University
Locations (1):
- Gaziantep Islam Science and Technology University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No